CLINICAL TRIAL: NCT00657878
Title: Liposomal Doxorubicin Versus Carboplatin/Paclitaxel in Patients With Ovarian Cancer Recurrence Between 6 and 12 Months After Previous Platinum Based Therapy: Phase III Randomized Multicenter Study Amendment Title Protocol Version 2.0: Phase III International Multicenter Randomized Study Testing the Effect on Survival of Prolonging Platinum-free Interval in Patients With Ovarian Cancer Recurring Between 6 and 12 Months After Previous Platinum Based Chemotherapy.
Brief Title: Efficacy Study of Chemotherapy to Treat Ovarian Cancer Recurrence by Prolonging the Platinum Free Interval
Acronym: MITO-8
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MITO-8; 2008-001755-22 (EudraCT Number)
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: platinum free interval; chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel; Topotecan; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- non platinum based chemotherapy (Experimental): a non platinum based therapy (corresponding to stealth liposomal doxorubicin, or topotecan, or gemcitabine,or any other drug approved in clinical practice for the treatment of patients with ovarian cancer after previous platinum-based chemotherapy) followed by a platinum based chemotherapy at disease progression
  Interventions: Drug: stealth liposomal doxorubicin; Drug: carboplatin; Drug: paclitaxel; Drug: Topotecan; Drug: Gemcitabine
- platinum based chemotherapy (Active Comparator): platinum based chemotherapy (corresponding to the combination of carboplatin + paclitaxel, or carboplatin + gemcitabine for patients with significant but lower than grade 3 neuropathy at baseline) followed by a non platinum based chemotherapy at disease progression
  Interventions: Drug: stealth liposomal doxorubicin; Drug: carboplatin; Drug: paclitaxel; Drug: Topotecan; Drug: Gemcitabine

INTERVENTIONS:
Drug: stealth liposomal doxorubicin — stealth liposomal doxorubicin 40 mg/m2 IV day 1 every 28 days
Drug: carboplatin — carboplatin AUC 5 IV day 1 every 21 days
Drug: paclitaxel — paclitaxel 175 mg/m2 IV day 1 every 21 days
Drug: Topotecan — dosing and schedule according to Institutional guidelines
Drug: Gemcitabine — 1000 mg/m2 on days 1,8,15 every 28 days

SUMMARY:
This study aims to test the hypothesis that the artificial prolongation of the platinum-free interval with a non-platinum treatment will improve the effectiveness of overall therapy in patients with ovarian cancer progression occurring 6-12 months after first-line treatment with a platinum-derivative.

DETAILED DESCRIPTION:
Ovarian cancer is the most deadly gynecologic cancer. Though many patients respond well initially to chemotherapy, most of them in time will suffer a relapse. Patients often receive multiple lines of chemotherapy for their recurrences, and the choice of chemotherapy depends largely on the time interval since the last therapy. Patients whose disease recurs longer than 12 months after a platinum containing treatment are considered to be platinum sensitive, and are candidates for retreatment with a platinum regimen.

Patients in whom disease recurs less than 6 months after a platinum containing treatment are considered platinum resistant or refractory, and are treated with a non platinum chemotherapy. The option of treatment is less clear for patients whose disease recurs between 6 and 12 months after platinum containing therapy. It is hypothesized that prolonging the interval since last platinum treatment by using a non platinum chemotherapy will result in better outcomes for these patients.

This study will evaluate if the experimental sequence of a non platinum based chemotherapy, followed at a later progression by a platinum based chemotherapy is superior, in terms of the effect on overall survival, to the standard inverse sequence of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of ovarian cancer
* Disease recurrence between 6 and 12 months after a first-line platinum based therapy
* Indication for chemotherapy, but no more than 2 previous lines of previous therapy
* Life expectancy of more than 3 months

Exclusion Criteria:

* Previous or concomitant malignant malignancy (excluding adequately treated baso-or squamocellular carcinoma of the skin and carcinoma in situ of the cervix)
* ECOG Performance Status at least 3
* Previous treatment with stealth liposomal doxorubicin
* Residual peripheral neuropathy Grade 3 or higher
* Heart disease (congestive heart failure, myocardial infarction within 6 months from study entry, atrioventricular block of any grade, severe arrhythmias)
* Neutrophils < 2000 x mm3, platelets < 100000 x mm3
* Inadequate renal function (creatinine no greater than 1.25 x normal values) or liver function (ALT or AST no greater than 1.25 x normal values)
* Present or suspected hemorrhagic syndromes
* Inability to comply with protocol and follow-up
* Inability to access study site for clinical visits
* Refusal of informed consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2008-11; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 18 months

SECONDARY OUTCOMES:
progression free survival | 18 months
changes in quality of life | 9 months
  quality of life is measured at baseline and at 3 months and 6 months after patient begins study
number of objective responses | 6 months
worst grade toxicity for each patient | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D., Principal Investigator — National Cancer Institute, Naples; Marilina Piccirillo, M.D., Principal Investigator — National Cancer Institute, Naples; Ciro Gallo, M.D., Ph.D., Principal Investigator — University of Campania Luigi Vanvitelli
Locations (40):
- Belgium (5):
  - AZ Groeninge, Kortrijk
  - UZ Gasthusiberg, Leuven
  - CHC-Clinique St-Joseph, Liège
  - Clinique & Maternité Sainte-Elisabeth, Namur
  - AZ Nikolaas, Sint-Niklaas
- Germany (8):
  - Charité Campus Virchow-Klinkum, Berlin
  - Kliniken essen Mitte-Evang Huyssens Stiftung/Knappschaft, Essen
  - Universitatsklinikum, Essen
  - Universitatsklinikum, Freiburg im Breisgau
  - Gynecology, Albertinen Krankenhaus, Hamburg
  - Universitatskilinikum Schleswig-Holstein, Kiel
  - Frauenklinik, Marburg
  - Klinikum rechts der Isar der Technischen Universitat, München
- Italy (27):
  - Azienda Ospedaliera V. Cervello, Palermo, PA
  - Ospedale S. Massimo, Day Hospital Oncologico, Penne, PE
  - Centro di Riferimento Oncologico, Divisione di Oncolgia Medica C, Aviano, PN
  - Ospedale Mazzoni, Ascoli Piceno
  - Policlinico Universitario, Bari
  - Universita di Bari Policinico I Clinical Ostetrica e Ginecologica, Bari
  - Ospedale Fatebenefratelli, Benevento
  - Ospedale Senatore Antonio Perrino, Brindisi
  - Universita Cattolica del Sacro Cuore, Campobasso
  - Ospedale Renzetti di Lanciano, Lanciano
  - Ospedale A. Manzoni, Lecco
  - Istituto Romagnolo per lo Studio e la Cura dei Tumori, Meldola
  - Istituto Europeo di Oncologia, Milan
  - Ospedale San Raffaele, Milan
  - Ospedale S. Gerardo, Monza
  - Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Uro-Ginecologico, Napoli
  - Ospedale Silvestrini, Perugia
  - Ospedale Civile S. Spirito, Pescara
  - A.O. Bianchi Melacrino Morelli Ospedale Riuniti, Reggio Calabria
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale degli Infermi, U.O. Oncologia Medica, Rimini
  - Ospedale S. Giovanni Calibita Fatebenefratelli, UO di Oncologia, Roma
  - Universita Cattolica del Sacro Cuore, Roma
  - A.O. Ordine Mauriziano, Torino
  - Ospedale S. Chiara, Trento
  - A.O. di Udine S. Maria della Misericordia, Udine
  - Ospedale Del Ponte, Varese

REFERENCES:
- [Derived] Piccirillo MC, Scambia G, Bologna A, Signoriello S, Vergote I, Baumann K, Lorusso D, Murgia V, Sorio R, Ferrandina G, Sacco C, Cormio G, Breda E, Cinieri S, Natale D, Mangili G, Pisano C, Cecere SC, Di Napoli M, Salutari V, Raspagliesi F, Arenare L, Bergamini A, Bryce J, Daniele G, Gallo C, Pignata S, Perrone F. Quality-of-life analysis of the MITO-8, MaNGO, BGOG-Ov1, AGO-Ovar2.16, ENGOT-Ov1, GCIG study comparing platinum-based versus non-platinum-based chemotherapy in patients with partially platinum-sensitive recurrent ovarian cancer. Ann Oncol. 2018 May 1;29(5):1189-1194. doi: 10.1093/annonc/mdy062. PMID 29462248